CLINICAL TRIAL: NCT03009838
Title: Letrozole Versus Laparoscopic Ovarian Drilling for Clomiphene-resistant Women With Polycystic Ovary Syndrome
Brief Title: Letrozole Versus Laparoscopic Ovarian Drilling in Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr., Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEVOD
Record Dates: First submitted 2017-01-01; First posted 2017-01-04 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- letrozole (Active Comparator): letrozole 2.5 mg oral tablets will be started daily from day 3 of the menses for 5 days in a dose of 5 mg/day
  Interventions: Drug: Letrozole
- laparoscopic drilling (Active Comparator): laparoscopy will be performed using three-puncture technique. Each ovary will be cauterized at four points, each for 4 seconds at 40 W for a depth of 4 mm with a mixed current, using a monopolar electrosurgical needle
  Interventions: Procedure: ovarian drilling

INTERVENTIONS:
Drug: Letrozole — oral tablets 2.5 mg
  Other Names: femara
  Arms: letrozole
Procedure: ovarian drilling — laparoscopic electrocauterization
  Arms: laparoscopic drilling

SUMMARY:
Polycystic ovary syndrome is the major cause of anovulatory infertility. Clomiphene citrate is the most commonly used oral agent for ovulation induction in this group, but there are some drawbacks with the use of it.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one year of infertility either primary or secondary.
* Body mass index: 25-35
* Normal fallopian tubes
* Normal semen analysis of the husband
* Women who will accept to participate in the study

Exclusion Criteria:

* Body mass index above 35
* Contraindication to general anesthesia
* Previous laparoscopic drilling
* Presence of other causes of infertility
* Women who had received metformin, gonadotrophin, oral contraceptives or other hormonal drugs during the preceding 6 months
* Women who intended to start a diet program
* Women who will refuse to participate in the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-01-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
The ovulation rate | 3 months

SECONDARY OUTCOMES:
The mid-cyclic endometrial thickness | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Franik S, Le QK, Kremer JA, Kiesel L, Farquhar C. Aromatase inhibitors (letrozole) for ovulation induction in infertile women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2022 Sep 27;9(9):CD010287. doi: 10.1002/14651858.CD010287.pub4. PMID 36165742